CLINICAL TRIAL: NCT03667664
Title: Prevention Study on Loss of Autonomy and Physical Dependence, Based on Physical Exercises and Nutrition Counseling Applied to Old People.
Brief Title: PREPA PREvention of Loss of Autonomy
Acronym: PREPA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL16_0324
Record Dates: First submitted 2018-01-29; First posted 2018-09-12 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-06

CONDITIONS: Mobility Limitation; Physical Activity
Keywords: Autonomy; Elderly; Physical exercise; Nutrition; Prevention
MeSH Terms: conditions — Mobility Limitation; Motor Activity | interventions — Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multicomponent group-based supervised exercise program (Other): Community-dwelling older adults aged of >70y, screened at risk of mobility disability risk factors and assessed with at least 1 mobility disability risk factor (see intervention 1). These subjects are included in the protocol and participate in a multicomponent exercise program.
  Interventions: Diagnostic Test: Multidimensional assessments; Other: Multicomponent group-based and supervised exercise program; Other: Follow-up at T3 + 6 months and T3 + 12 months

INTERVENTIONS:
Diagnostic Test: Multidimensional assessments — Evaluation carried out during a day hospital at T0 (initial assessment) and T3 following the exercise program including:
  1. Clinical assessment by a geriatrician
  2. Nutritional assessment
  3. Physical capacity assessment
  Following initial assessment (T0), older adults are included in the multicomponent exercise program if they present mobility disability risk factors including :
  * At least pre-frailty regarding Fried frailty criteria AND/OR
  * At least probable sarcopenia regarding EWGSOP2 algorithm AND/OR
  * The presence of at least an intermediate fall risk AND/OR
  * The presence of a fear of falling Following the exercise program (T3), all participants are re-assessed in the same way as T0. Investigators then set goals in physical activity with participants to maintain benefits and foster self-engagement in an healthy lifestyle. Additionnally, participants are orientated to exercise facilities and received an individualized booklet of exercises for home-based training.
Other: Multicomponent group-based and supervised exercise program — The intervention consists in a progressive multicomponent exercise training protocol. There are 2 sessions per week of 1 hour each for a total of 12 weeks. Sessions involve functional, resistance and balance exercises. Intensity is based on rating perceived effort (Borg's scale CR1-10) and volume towards 1 to 3 sets of 6 to 15 repetitions. Progressiveness in intensity and volume was based on effort tolerance, contraction regimen, velocity and load. Training schedule is described elsewhere (Delaire et al, 2023 ; doi.org/10.3390/nu15194100). Participants are allocated to an homogenous group based on functional status and cardiorespiratory comorbidities. Trained kinesiologists supervised the exercise program. Participants used free weights and elastic bands.
Other: Follow-up at T3 + 6 months and T3 + 12 months — Follow-up at T3+6 months:
  Investigators interviewed participants for 30 minutes. During the interview, data collection include:record of undesirable events in the interval T3 / T3+6 (falls, unscheduled hospitalization, illness, institutionalization), medication changes, ADL, IADL, FES-I, and RAPA. Goal-settings at T3 are adjusted if not reach. Finally, investigators stimulate intrinsic motivation for PA.
  Follow-up at T3 + 12 months:
  Investigators re-assessed physical capacity, physical activity level, quality of life, fall risk and frailty for the last visit. Data collection include:
  * SPPB
  * Handgrip test and maximal isometric strength of the quadriceps
  * Questionnaires : SarQoL©, FES-I, RAPA
  * Gait quality analysis using inertial sensors
  * Undesirable events in the interval T3+6 / T3+12 (falls, unscheduled hospitalization, illness, institutionalization)
  * Medication changes
  * Body mass index
  * ADL and IADL At last, goals in physical activity are adjusted if they are still not reach

SUMMARY:
According to several reports, the proportion of people aged 80yrs or older will be doubled within the next 25y, reaching 10% of the global population. Furthermore, the health life expectancy at 65y is 10.4y which remains much lower than the general life expectancy. As a result, there is a constant need of developing preventive strategies through multimodal programs.

Among the predictive factors of mobility disability with age, muscular weakness and decreased physical function are major components. These two factors are known of being responsible for falls and fractures that lead to decrease the quality of life and an increase in mortality.

Exercise and nutrition are the only components that have proven their efficacy to struggle mobility disability risk. It is important to integrate these two components in a sustained intervention within a multidimensional prevention program. However, there is a lack of implementation of these programs in primary care.

Indeed, neither the screening of older adults at risk of mobility disability, nor the preventive actions are usually implemented for this population. The implementation of a prevention care pathway, with personalized intervention and a sustained follow-up, along with supervised exercise training combined with nutritional counselling, is the public health imperatives.

Based on prevention care pathway that designed for community-dwelling older adults screened at risk of mobility disability. The purpose of this open cohort study was to highlight the efficacy and the feasibility of a multimodal program implemented on real-life setting specifically on the physical function and risk of mobility loss, along with their maintenance at 6-months and 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for the "mobility loss prevention" program
* At least one of the following signs:

  * Difficulty carrying a loaded shopping basket (about 4.5 kg)
  * Difficulty rising from a chair without using the arms
  * Difficulty climbing one flight of stairs (10 steps)
  * Difficulty moving around
  * Slowed walking
  * Difficulty walking more than 400 meters without stopping
  * Walking time < 30 minutes/day
  * Fatigue during mild physical efforts: running errands, household chores; fear of falling and/or at least one fall in the past year
  * Recent unintentional weight loss: weight loss ≥ 5% in 6 months or BMI < 22 kg/m²

Exclusion Criteria:

* Patient who has not given consent to participate
* Patient under guardianship in retrospective phase
* Locomotor disability
* expectancy of life being under 12 months
* BMI ≥ 35 Kg/m2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Functional status | initial assessment (baseline), following the exercise program (month 3), last visit (month 15)
  Functional status is assessed using the overall SPPB (Short Physical Performance Battery) score based on three components: 6 meters usual walking speed, 5 repetitions chair stand test, and static balance tests. (composite score /12). The SPPB score is calculate from the results in 3 subtests. It ranges from 1 to 12 points. Clinically meaningful change is 1 point.

SECONDARY OUTCOMES:
Evaluation of effectiveness on muscle strength : Handgrip test (kg) | initial assessment (baseline), following the exercise program (month 3), last visit (month 15)
  The subject has to perform 3 maximum isometric contractions on a dynamometer which records the force developed. The average of these 3 values will be retained. A value lower than <16kg for women and <27kg for men are considered abnormal and indicate the presence of probable sarcopenia.
Evaluation of effectiveness on muscle strength : Maximal isometric strength of the quadriceps (kg) | initial assessment (baseline), following the exercise program (month 3), last visit (month 15)
  The subject has to perform 3 maximum isometric muscular contractions separately against a dynamometer. The best performance (i.e. greatest strength measure) is collected.
Evaluation of effectiveness on functional status : 5 repetitions chair stand test (s) | initial assessment (baseline), following the exercise program (month 3), last visit (month 15)
  The subject has to stand with knee extended and sit from a chair 5 times without stopping
Evaluation of effectiveness on functional status : Time in TUG (s) | initial assessment (baseline), following the exercise program (month 3), last visit (month 15)
  The subject must get up from a chair, walk at usual speed 3 meters, turn around, and sit down again. A value greater than or equal to 20 seconds will be considered abnormal.
Evaluation of effectiveness on functional status : Lower body muscle power measured by a one sit-to-stand test perform at maximum speed (Neurocom Balance Master, Medimex®, France) | initial assessment (baseline), following the exercise program (month 3)
  Estimation of lower limb muscle power based on the mean of the 3 repetitions of a sit-to-stand test perform separately. For each transfer, the lifting index (as a % of body weight), reaction time (s), the oscillation limit of the center of gravity, and the symmetry of the supports are measured
Evaluation of effectiveness on functional status : Gait quality analysis using inertial sensors (GaitUp, MindMaze®, Switzerland) | initial assessment (baseline), following the exercise program (month 3), last visit (month 15)
  A 50 meters walking test perform at usual speed is realized. Data collection include : gait speed, gait variability, gait asymmetry, % flight time, % support time, % double support time, angle of attack, push-off angle, step height, step length, number of cycles in the U-turn, angles in the U-turn
Evaluation of muscle mass : SMI measured by bio-impedance analysis (kg.m2) | initial assessment (baseline), following the exercise program (month 3)
  SMI is a relative index which is computed from the Sergi equation. Cut-off points are <7,0 and <5,5 for men and women respectively and are considered abnormal. These are the reference values for sarcopenia diagnosis.
Evaluation of muscle mass : Ultrasonography of the vastus lateralis | initial assessment (baseline), following the exercise program (month 3)
  Data collection of muscle density (cm)
Evaluation of muscle mass : Ultrasonography of the vastus lateralis | initial assessment (baseline), following the exercise program (month 3)
  Data collection include of pennation angle (degree)
Evaluation of muscle mass : Ultrasonography of the vastus lateralis | initial assessment (baseline), following the exercise program (month 3)
  Data collection include of fiber length (cm)
Evaluation of dependencies : Katz scale (Activities of Daily Living - ADL) | initial assessment (baseline), following the exercise program (month 3), last visit (month 15)
  Katz scale (ADL) consists of 6 questions. Score varies from 0 to 6. The lower the score, the more dependant is the patient
Evaluation of dependencies : Lawton scale (Instrumental Activities of Daily Living-IADL) | initial assessment (baseline), following the exercise program (month 3), last visit (month 15)
  Lawton scale (IADL) consists of 8 questions. Score varies from 0 to 8. The lower the score, the more dependant is the patient.
Record of undesirable events : Falls, unscheduled hospitalization, illness, institutionalization | initial assessment (baseline), following the exercise program (month 3), 6 months following the exercise program (month 9), last visit (month 15)
  Data are collected between intervals :
  T3/T3+6 and T3+6/T3+12
Evaluation of fear of falling : FES-I questionnaire (/64) | initial assessment (baseline), following the exercise program (month 3), last visit (month 15)
  The validated French translated form is used. Questionnaire is self-administrated.
  FES-I questionnaire (Falls Efficacy Scale-International) consists of 16 questions. Score varies from 16 to 64.
  A fear of falling is considered to be present with score >23.
Evolution of the level of physical activity : RAPA questionnaire (/10) | initial assessment (baseline), following the exercise program (month 3), last visit (month 15)
  The RAPA is validated physical activity questionnaire in older adults. The score is calculated from the reported information of each visit.
  Score varies from 0 to 10. The higher the score, the more physically active is the patient.
Evolution of quality of life : SarQoL© questionnaire | initial assessment (baseline), following the exercise program (month 3), last visit (month 15)
  The SarQoL© is a validated questionnaire in sarcopenic older adults. French validated translated form were used. The questionnaire is self-administrated. An overall change of 7,35 points in the questionnaire is considered to be clinically meaningful.
Evaluation of biomarkers : risk of fractures - Calcemia (mmol/L) | initial assessment (baseline), following the exercise program (month 3)
  initial assessment (baseline), following the exercise program (month 3)
Evaluation of biomarkers : risk of fractures - Vitamin D (nmol/L). | initial assessment (baseline), following the exercise program (month 3)
  initial assessment (baseline), following the exercise program (month 3)
Evaluation of biomarkers : exploratory Fibroblast Growth Factor 19 (FGF-19) (pg/L) | initial assessment (baseline), following the exercise program (month 3)
  FGF-19 is analysed in plasma samples by ELISA method. Blood sample is collected in routine care.
Evaluation of biomarkers : nutritional status - Albumin (g/L) | initial assessment (baseline), following the exercise program (month 3)
  Albumin (g/L)
Evaluation of biomarkers : nutritional status - Pre-albumin (g/L) | initial assessment (baseline), following the exercise program (month 3)
  Pre-albumin (g/L)
Evaluation of biomarkers : inflammation C-reactive protein | initial assessment (baseline), following the exercise program (month 3)
Evaluation of physical frailty : Fried criteria | initial assessment (baseline), following the exercise program (month 3), last visit (month 15)
  Fried criteria include : unvolontary weight loss >5% during the last 12 months, self-reported exhaustion, low gait speed, low grip strength and poor physical activity level. 0 criterion = non frail ; 1-2 criteria = pre-frail ; ≥3 criteria = frail
Evaluation of sarcopenia : EWGSOP2 | initial assessment (baseline), following the exercise program (month 3)
  No sarcopenia = muscle strength and mass normal Probable sarcopenia = low muscle strength, normal muscle mass Sarcopenia = low muscle strength and mass Severe sarcopenia = low muscle strength and mass + poor physical performances
Evaluation of nutritional status : Mini Nutritional Assessment | initial assessment (baseline), following the exercise program (month 3)
  This self-administrated questionnaire consists of 18 questions. Score varies from 0 to 30. From 17 to 24 points : risk of malnutrition Less than 17 points : poor nutritional status
Evaluation of nutritional status : caloric (kcal) needs and intakes from the dietary survey | initial assessment (baseline), following the exercise program (month 3)
  Survey is self-administrated. Needs/Intake are calculated based on the survey.
Evaluation of nutritional status : protein (g/J) needs and intakes from the dietary survey | initial assessment (baseline), following the exercise program (month 3)
  Survey is self-administrated. Needs/Intake are calculated based on the survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Gériatrique Groupement Hospitalier Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No